CLINICAL TRIAL: NCT02781402
Title: Relationship Between Body Mass Index and Heart Rate Recovery Following 4 Weeks of Aerobic Training Among Young Physically Inactive Adults
Brief Title: Relationship Between BMI & HRR After 4 Weeks of Aerobic Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Mr, Universiti Tunku Abdul Rahman
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/SERC/82/2015
Record Dates: First submitted 2016-05-13; First posted 2016-05-24 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Overweight
Keywords: Overweight BMI Individuals; Normal BMI Individuals; Recovery Heart Rate
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Same intervention (4 weeks of aerobic training) was given to 2 different groups (Normal BMI group & Overweight BMI group).
Who Masked: Outcomes Assessor
Masking Description: Assessor who measured pre and post outcomes was blended and did not know participants belonged to which group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4 weeks of Aerobic Training for normal BMI group (Experimental): 4 weeks of aerobic training on treadmill 3 times per week.
  Interventions: Procedure: 4 weeks of Aerobic Training
- 4 weeks of Aerobic Training for overweight BMI group (Experimental): 4 weeks of aerobic training on treadmill 3 times per week.
  Interventions: Procedure: 4 weeks of Aerobic Training

INTERVENTIONS:
Procedure: 4 weeks of Aerobic Training — The duration of aerobic training was 40 minutes for each session and 3 days per week with the intensity of 75-80% of their maximum heart rate. The participants were needed to walk or jog on treadmill during the first 10 minutes at the intensity of 50-60% of maximal heart rate (HR max). The aerobic training was followed by 4 x 4 minutes intervals at 75-80% HR max. The participants were given 3 minutes active breaks in between the intervals in which they can either walk or jog at 50-60% of maximal heart rate.

SUMMARY:
World Health Organization (WHO) defined body mass index (BMI) as the ratio of weight in kilograms to the square of the height in meters (kg/m2). BMI has been used widely to diagnose obesity as it is a simple method to be carried out and is also inexpensive. According to WHO, there were 1.9 billion overweight individuals in 2014 with the age of 18 years old or above. Of 1.9 billion overweight individuals, there were 600 million obese adults. The prevalence of cardiovascular disease is higher among the overweight and obese individuals compared to individuals with normal body mass index. This probably is due to altered cardiovascular autonomic regulation. The risk of getting cardiovascular diseases is also higher among physically inactive individuals. As much as 60% of American adults are not regularly active and 25% of them are not active at all. Obese and overweight individuals tend to be physically inactive and it has been shown that there is a negative relationship between BMI and heart rate recovery (HRR). HRR is defined as difference in heart rate between maximum exercise and 1 minute later during recovery period after stopping of exercise. HRR after exercise stress is due to withdrawal of sympathetic nervous system and the reactivation of parasympathetic nervous system. Parasympathetic nervous system is altered in obese individuals therefore leading to poor HRR after exercise. Aerobic training not only can reduce the body composition but also improves the autonomic cardiovascular control. There is limited literature support for any study which shows that potential of 4 weeks aerobic training can influence the heart rate recovery in sedentary healthy adults. Most of studies conducted were using minimum of 6 to 8 weeks of aerobic training. The potential of 4 weeks of aerobic training in improving the autonomic nervous system among sedentary adults is still unclear. Therefore, we hypothesized in our study that there will be effect of 4 weeks of aerobic training on vagal modulation.

DETAILED DESCRIPTION:
Obesity is a complex health issue that results from various causes and contributing factors. Individual factors like genetics and behavior may contribute to overweight and obesity. Genetics played an important role in increasing hunger and food intake of individuals. A few examples of common diseases that are related to obesity are type-2 diabetes, stroke, coronary heart disease and some types of cancer. All these obesity related diseases may not be fully reversible even after weight loss . Body mass index (BMI) is used widely as a screening tool to assess overweight and obesity. Based on the World Health Organization (WHO) international classification of BMI, individuals are considered as obese if their BMI value is equal to 30 kg/m2 or higher and overweight if BMI is 25-29.9 kg/m2. A study was conducted in USA to find the prevalence of obesity among children and adults. Researchers attempted to predict the childhood obesity and analyse the obesity trend among adults in United States. The results of the study showed that the prevalence of obesity among children were 16.9% and adults were 34.9%. There were no obvious changes in prevalence of obesity among children and adults in between 2003-2012 in United States (1). It cannot be denied that there is a link between increasing rate of obesity and increasing medical spending. Medical spending for obese individuals was 42% higher compared to those with normal body weight (2). The researchers reported in their study that obesity was one of the factors that became an economic burden for both public and private payers. South East Asia and Western Pacific countries suffer from diseases associated with obesity such as cardiovascular diseases and diabetes. Malaysia is the country the highest rate of obesity in South East Asia (3). Studies have showed that autonomic nervous system is associated with obesity. In 2001, a study was conducted to identify the effect of weight loss on autonomic nervous system. The findings showed that the activity of parasympathetic nervous system increased with weight loss and cardiac vagal tone improved significantly after weight loss (4). Cardiac vagal tone is controlled mainly by parasympathetic nervous system and this helps to improve the heart rate recovery (HRR). There are two phase of heart rate recovery, fast and slow phase. The fast phase is due to cardiac parasympathetic reactivation while the slow phase is because of cardiac sympathetic withdrawal. If there is any disturbance of the autonomic nervous system then the HRR will slow down (5). Therefore, HRR can be used to assess the cardiac autonomic function and as a marker of cardiac vagal tone. Abnormal heart rate recovery after exercise stress can be considered as dysfunction of autonomic nervous system. It has been suggested in several studies that heart rate recovery after exercise stress is slower among obese individuals compared to BMI individuals. A study was conducted to identify the relationship between heart rate recovery and body mass index. The finding showed that there was a negative association between heart rate recovery and body mass index. 3.5% of 2443 individuals presented with delayed decrease heart rate recovery. The prevalence of decreased heart rate recovery was higher among overweight and obese groups (6). In another study similar findings were observed. Researchers concluded that obese individuals are more likely to have an impaired heart rate recovery during the recovery phase after exercise (7). Aerobic training improves the autonomic cardiovascular control. A study on 4 weeks of aerobic training was done to identify its effects on cardiac vagal tone. Authors reported that 4 weeks of treadmill aerobic training was able to improve the autonomic nervous system among pre-hypertension individuals (8). The aerobic training consisted of 30 minutes treadmill exercise at 65% of maximum oxygen consumption. Another study showed the similar results in which the autonomic nervous system was improved after 6 months of moderate intensity aerobic training (9). The aerobic training was carried out 1 hour each session with 2 sessions in one week for 6 months. The present systematic review shows that aerobic training has been proven to be effective in increasing the heart rate recovery among subjects with established heart disease (10). The effects of 4 weeks of aerobic training in improving the cardiac vagal tone among sedentary healthy adults are still unclear. Therefore, we aim to study the effects of 4 weeks of aerobic training on vagal modulation.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary subjects
2. Age between 18 to 25 years old
3. Body mass index range = 18.50 - 24.9 kg/m² (normal) = 25 - 29.9 kg/m² (overweight)

Exclusion Criteria:

1. Subjects with cardiovascular disease
2. Subjects with musculoskeletal problem
3. Not willing to participate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Recovery | At baseline and After 4 weeks of aerobic training
  The participants were required to take part in the exercise testing before beginning the 4 weeks of aerobic training. Ebbeling submaximal treadmill (EbbTM) protocol was used during the exercise testing. Finger pulse oximeter was placed on the participants' finger. The particiapnts were required to warm up for 4 minutes by walking at the speed that maintains the heart rate within 50% to 70% of their maximum heart rate (HR max) without any inclination (0% grade). Following 4 minutes of warm up, the participants walked at the same speed for another 4 minutes at a grade of 5%. After cessation of exercise test, heart rate was immediately recorded from the pulse oximeter for 1 minute. The heart rate was measured during the passive recovery phase in which the participants were in supine position.

SECONDARY OUTCOMES:
Change in Body Mass Index | At baseline and After 4 weeks of aerobic training
  BMI to be measure before and at end of 4 weeks of aerobic training to see any differences and impact of aerobic training on BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Imtiyaz Ali Mir, Principal Investigator — Universiti Tunku Abdul Rahman

IPD SHARING:
Plan to Share IPD: No
Confidentiality of participants.

REFERENCES:
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Rissanen P, Franssila-Kallunki A, Rissanen A. Cardiac parasympathetic activity is increased by weight loss in healthy obese women. Obes Res. 2001 Oct;9(10):637-43. doi: 10.1038/oby.2001.84. PMID 11595781
- [Background] Brinkworth GD, Noakes M, Buckley JD, Clifton PM. Weight loss improves heart rate recovery in overweight and obese men with features of the metabolic syndrome. Am Heart J. 2006 Oct;152(4):693.e1-6. doi: 10.1016/j.ahj.2006.07.019. PMID 16996838
- [Background] Barbosa Lins TC, Valente LM, Sobral Filho DC, Barbosa e Silva O. Relation between heart rate recovery after exercise testing and body mass index. Rev Port Cardiol. 2015 Jan;34(1):27-33. doi: 10.1016/j.repc.2014.07.006. Epub 2015 Jan 8. English, Portuguese. PMID 25577658
- [Background] Gondoni LA, Titon AM, Nibbio F, Augello G, Caetani G, Liuzzi A. Heart rate behavior during an exercise stress test in obese patients. Nutr Metab Cardiovasc Dis. 2009 Mar;19(3):170-6. doi: 10.1016/j.numecd.2008.07.001. Epub 2008 Sep 19. PMID 18804987
- [Background] Collier SR, Kanaley JA, Carhart R Jr, Frechette V, Tobin MM, Bennett N, Luckenbaugh AN, Fernhall B. Cardiac autonomic function and baroreflex changes following 4 weeks of resistance versus aerobic training in individuals with pre-hypertension. Acta Physiol (Oxf). 2009 Mar;195(3):339-48. doi: 10.1111/j.1748-1716.2008.01897.x. Epub 2008 Sep 4. PMID 18774947
- [Background] Gulli G, Cevese A, Cappelletto P, Gasparini G, Schena F. Moderate aerobic training improves autonomic cardiovascular control in older women. Clin Auton Res. 2003 Jun;13(3):196-202. doi: 10.1007/s10286-003-0090-x. PMID 12822041
- [Background] Snoek JA, van Berkel S, van Meeteren N, Backx FJ, Daanen HA. Effect of aerobic training on heart rate recovery in patients with established heart disease; a systematic review. PLoS One. 2013 Dec 18;8(12):e83907. doi: 10.1371/journal.pone.0083907. eCollection 2013. PMID 24367618
- [Result] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244